CLINICAL TRIAL: NCT02633189
Title: A Randomized Open-label Phase 3 Trial Comparing Bevacizumab + Erlotinib vs Erlotinib Alone as First Line Treatment of Patients With EGFR Mutated Advanced Non Squamous Non Small Cell Lung Cancer
Brief Title: Study Comparing Bevacizumab + Erlotinib vs Erlotinib Alone as First Line Treatment of Patients With EGFR Mutated Advanced Non Squamous Non Small Cell Lung Cancer
Acronym: BEVERLY
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BEVERLY; 2015-002235-17 (EudraCT Number)
Record Dates: First submitted 2015-12-15; First posted 2015-12-17 (Estimated); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Non-squamous Non-small Cell Lung Cancer
Keywords: stage IV; stage IIIB; EGFR mutation; non-squamous; liquid biopsy; erlotinib; bevacizumab
MeSH Terms: interventions — Erlotinib Hydrochloride; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- erlotinib and bevacizumab (Experimental)
  Interventions: Drug: Erlotinib; Drug: Bevacizumab
- erlotinib (Active Comparator)
  Interventions: Drug: Erlotinib

INTERVENTIONS:
Drug: Erlotinib — given orally 150 mg daily
Drug: Bevacizumab — 15 mg/kg intravenously every 21 days.
  Arms: erlotinib and bevacizumab

SUMMARY:
The purpose of this study is to test whether the combination of bevacizumab and erlotinib can prolong progression free survival as compared with erlotinib alone as first-line treatment in patients with non small cell lung cancer (NSCLC) with activating mutation of EGFR.

DETAILED DESCRIPTION:
The co-primary objectives are to assess investigator-assess, and blinded independent centrally-reviewed progression-free survival .

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Histological documentation of primary non squamous lung carcinoma
3. Stage IV or IIIB disease with supraclavicular metastatic nodes (according to TNM 7th edition)
4. Activating epidermal growth factor receptor mutation (exon19 deletion or exon 21 L858R mutation or other activating/sensitizing mutations, such as exon 21 L861Q, exon 18 G719S, G719A and G719C, exon 20 S768I and V769L). EGFR mutation testing must be performed at participating centres in a certified lab (AIOM-SIAPEC program or other European Quality Assurance [EQA] schemes)
5. Clinical or radiologic evidence of disease (at least one target or non target lesion according to RECIST 1.1)
6. ECOG performance status 0 to 2
7. Life expectancy > 3 months
8. Use of an acceptable mean of contraception for men and women of childbearing potential
9. Written informed consent.

Exclusion Criteria:

1. EGFR T790M mutation alone or exon 20 insertions as unique mutation
2. Tumors with a squamous component
3. Prior chemotherapy or any other medical treatment for advanced NSCLC (previous neoadjuvant or adjuvant chemotherapy is allowed if > 6 months before randomisation)
4. Radiotherapy to any site for any reason within 28 days prior to randomization (palliative radiotherapy to bone lesions is allowed if ≥ 14 days before randomization)
5. Full-dose anticoagulation with warfarin
6. Current or recent (within 10 days of enrolment) use of aspirin (>325 mg/day) or chronic use of other full-dose nonsteroidal anti-inflammatory drugs (NSAIDs) with anti-platelet activity
7. Receiving any medications or substances that are strong or moderate inhibitors of cytochrome P450 3A4 (CYP3A4) are prohibited =< 7 days prior to registration
8. Receiving any medications or substances that are inducers of CYP3A4 use of inducers are prohibited =< 7 days prior to registration
9. Inadequate coagulation parameters:

   * activated partial thromboplastin time (APTT) >1.5 x the upper limit of normal (ULN) or
   * INR >1.5
10. Inadequate liver function, defined as:

    * serum (total) bilirubin >1.5 x ULN
    * AST/SGOT or ALT/SGPT >2.5 x ULN
11. Inadequate renal function, defined as:

    * serum creatinine >2.0 mg/dl or >177 micromol/l
    * urine dipstick for proteinuria >2+. Patients with > o = 1+ proteinuria at baseline dipstick analysis must undergo a 24-hour urine collection and must demonstrate ≤1g of protein in their 24-hour urine collection.
12. Pregnancy or breast-feeding
13. Inadequately controlled hypertension (defined as systolic blood pressure >150 and/or diastolic blood pressure >100 mmHg on antihypertensive medications)
14. History of gross hemoptysis within 3 months prior to randomization unless definitively treated with surgery or radiation
15. History of any of the following within 6 months prior to randomisation: serious systemic disease, unstable angina, New York Heart Association (NYHA) Grade 2 or greater Congestive Heart Failure (CHF), unstable symptomatic arrhythmia requiring medication, clinically significant peripheral vascular disease, abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess
16. Serious, non-healing wound, ulcer, or bone fracture
17. Evidence of bleeding diathesis or coagulopathy or other serious or acute internal bleeding within 6 months prior to randomization
18. Central Nervous System (CNS) bleeding; history or clinical evidence of CNS stroke (hemorrhagic or thrombotic) within the last 6 months
19. In-patient surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to randomization
20. Minor surgical procedure, fine needle aspirations or core biopsy within 7 days prior to randomization
21. Anticipation of need for a major surgical procedure during the course of the study
22. Inability to take oral medication or requirement for intravenous (IV) alimentation or total parenteral nutrition with lipids, or prior surgical procedures affecting absorption
23. Evidence of confusion or disorientation, or history of major psychiatric illness that may impair the patient's understanding of the Informed Consent Form or his/her ability to comply with study requirements
24. Any other invasive malignancies within 5 years (except for adequately treated carcinoma in situ of the cervix or basal or squamous cell skin cancer or surgically resected prostate cancer with normal PSA)
25. Brain metastasis
26. Patients who have had radiotherapy ≥ 4 weeks prior to the first dose of study treatment, but who are still experiencing acute toxic effects of radiotherapy
27. Known HIV positive patients (patients with both acute or chronic infection are excluded)
28. Active HBV or HCV infection (patients with chronic non-active infection are eligible)
29. Any already known inflammatory changes of the surface of the eye at baseline
30. Any other concomitant pathologies or laboratory alterations that prevent or contraindicate the use of erlotinib or bevacizumab.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-04 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
progression free survival | up to 2 years
  as determined by investigator
progression free survival | up to 2 years
  as determined by an independent central review board blinded to study treatment

SECONDARY OUTCOMES:
overall survival | 1 year
changes in quality of life scores from baseline | up to 2 years
number of patients with complete and partial responses , investigator assessed | 6 months
number of patients with complete and partial responses , centrally reviewed | 6 months
worst grade toxicity per patient | up to one year
progression free survival according to type of EGFR mutation (exon 19del, exon 21L858R, other) | 2 years

OTHER OUTCOMES:
number and type of EGFR mutations in plasma samples | up to 2 years
  samples taken at baseline, 6 weeks, 6 months, and at progression

CONTACTS AND LOCATIONS:
Overall Officials: Cesare Gridelli, M.D., Principal Investigator — S.G.Moscati Hospital
Locations (55):
- Italy (55):
  - Ospedale Ramazzini, Day Hospital Oncologico, Carpi, MO
  - Casa di Cura La Maddalena S.p.A., Dipartimento Oncologico, Palermo, PA
  - Ospedale di Prato, Prato, PO
  - Ospedale S. Chiara, Trento, TN
  - Ospedale S. Bortolo ULSS 6, U.O. di Oncologia Medica, Vicenza, VI
  - A.S.O. SS Antonio e Biagio e Cesare Arrigo, Alessandria
  - A.O. S. Giuseppe Moscati, Avellino
  - Centro Riferimento Oncologico, Aviano
  - AO G. Rummo, Benevento
  - Ospedale Senatore Antonio Perrino, Brindisi
  - Ospedale A. cardarelli, Campobasso
  - U.L.S.S. 15 Veneto, Camposampiero
  - A.O. Garibaldi Nesima, Catania
  - Centro Clinico Diagnostico G.B. Morgagni, Catania
  - Policlinico vittorio Emanuele, Catania
  - Ospedale Civile per gli Infermi, Faenza
  - Ospedale S. Croce, Fano
  - A.O.U. Arcispedale Sant'Anna, Ferrara
  - Ospedale Villa Scassi, Genova
  - Ospedale di Guastalla, Guastalla
  - A.O. Vito Fazzi, Lecce
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola
  - Istituto Europeo di Oncologia, Milan
  - Istituto Nazionale Tumori, Milan
  - Ospedale San Paolo, Milan
  - A.O. U.L.S.S. 13, Mirano
  - A.O.U. Policlinico Modena, Modena
  - Azienda Ospedaliera Cardarelli, Napoli
  - A.O.U. Seconda Università di Napoli, Napoli
  - AORN Ospedale dei Colli - Osp Monaldi, Napoli
  - Istituto Nazionale Tumori Fondazione G. Pascale, Napoli
  - Istituto Sacro Cuore Don Calabria, Negrar
  - A.O.U. Maggiore della Carità, Novara
  - Istituto Oncologico Veneto, Padua
  - Policlinico Giaccone, Palermo
  - Fondazione Salvatore Maugeri, Pavia
  - Osp. S. Maria della Misericordia, Perugia
  - A.O. Ospedali Riuniti Marche Nord, Pesaro
  - Ospedale Guglielmo da Saliceto, Piacenza
  - A.O. San Carlo, Potenza
  - Ospedale Santa Maria delle Croci - AUSL, Ravenna
  - Ospedale Umberto I, Ravenna
  - Ospedale degli Infermi Rimini - Ospedale Cervesi Cattolica, Rimini
  - IRCCS Centro di Riferimento Oncologico Basilicata, Rionero in Vulture
  - Istituto Regina Elena, Roma
  - Ospedale Camillo Forlanini, Roma
  - Ospedale S. Giovanni Calibita Fatebenefratelli, Roma
  - Policlinico Universitario Campus Bio Medico, Roma
  - Ospedale di Sondrio, Sondrio
  - Ospedale Fabrizio Spaziani di Frosinone, Sora
  - Ospedale Maggiore, Trieste
  - Azienda Ospedaliero-Universitaria S.M. della Misericordia di Udine, Udine
  - Ospedale S. Andrea, Vercelli
  - A.O.U. Integrata, Verona
  - ASL Viterbo - Ospedale Belcolle, Viterbo

REFERENCES:
- [Derived] Piccirillo MC, Bonanno L, Garassino MC, Esposito G, Dazzi C, Cavanna L, Burgio MA, Rosetti F, Rizzato S, Morgillo F, Cinieri S, Veccia A, Papi M, Tonini G, Gebbia V, Ricciardi S, Pozzessere D, Ferro A, Proto C, Costanzo R, D'Arcangelo M, Proietto M, Gargiulo P, Di Liello R, Arenare L, De Marinis F, Crino L, Ciardiello F, Normanno N, Gallo C, Perrone F, Gridelli C, Morabito A. Addition of Bevacizumab to Erlotinib as First-Line Treatment of Patients With EGFR-Mutated Advanced Nonsquamous NSCLC: The BEVERLY Multicenter Randomized Phase 3 Trial. J Thorac Oncol. 2022 Sep;17(9):1086-1097. doi: 10.1016/j.jtho.2022.05.008. Epub 2022 Jun 1. PMID 35659580
- [Derived] Deng Z, Qin Y, Liu Y, Zhang Y, Lu Y. Role of Antiangiogenic Agents Combined With EGFR Tyrosine Kinase Inhibitors in Treatment-naive Lung Cancer: A Meta-Analysis. Clin Lung Cancer. 2021 Jan;22(1):e70-e83. doi: 10.1016/j.cllc.2020.08.005. Epub 2020 Sep 18. PMID 33067126